CLINICAL TRIAL: NCT05373784
Title: Outcomes of Fecal Microbiota Transplantation (FMT) in Uncomplicated Diverticulitis: A Pilot Study
Brief Title: FMT in Uncomplicated Diverticulitis
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Justin Maykel (Other)
Responsible Party: Sponsor-Investigator, Justin Maykel, Professor of Surgery, University of Massachusetts, Worcester
Organization: University of Massachusetts, Worcester (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000055
Record Dates: First submitted 2022-05-09; First posted 2022-05-13 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: Diverticulitis; Uncomplicated Diverticular Disease
MeSH Terms: conditions — Diverticulitis | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: This will be a pilot study of 10 patients with a diagnosis of uncomplicated diverticulitis who will undergo FMT.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- FMT cohort (Experimental): This will be a single-arm pilot study of patients with uncomplicated diverticulitis. All subjects enrolled as recipients will undergo FMT via colonoscopy.
  Interventions: Biological: Fecal Microbiota Transplantation (FMT)

INTERVENTIONS:
Biological: Fecal Microbiota Transplantation (FMT) — Fecal microbiota transplantation (FMT) involves administering fecal material from a healthy individual into the gastrointestinal tract of another individual. This is currently an accepted method of treatment for recurrent colitis secondary to Clostridium difficile infection refractory to antibiotics/medical management. FMT can be delivered via capsule endoscopy or via colonoscopy. In this study, it will be administered via colonoscopy.

SUMMARY:
Fecal Microbiota Transplantation (FMT) is an established treatment for Clostridium difficile (C. diff) infection refractory to medical management. As C. diff infection usually arises due to significant disturbances in the gut microbiome, FMT is typically performed to restore a healthy microbiome among affected patients who have failed other treatments. Diverticulitis is a major, and often recurrent, source of morbidity in the U.S for which antibiotics and surgical resection constitute the only treatment options to date. Although alterations of the intestinal microbiome have also been shown among patients with diverticular disease, research on FMT in diverticulitis is sparse. The intended goal of this project is to determine the feasibility, effectiveness and safety of FMT in the treatment of uncomplicated diverticulitis, using clinical outcomes and microbiome analyses.

DETAILED DESCRIPTION:
This study aims to assess the safety and efficacy of fecal microbiota transplantation (FMT) in treating uncomplicated diverticulitis. FMT will be delivered via colonoscopy using donor stool. Fecal material samples obtained from the University of Minnesota Microbiota Therapeutics Program (UMMTP) will be used each patients FMT. These samples undergo FDA mandated testing prior to being used as donor samples.

Recipients will undergo FMT via Colonoscopy at UMASS Memorial Medical Center and will be monitored for one hour after the procedure to ensure they are not experiencing any adverse events. They will receive a phone call 24 hours and 2 weeks after their procedure to ensure that they are at their baseline health. Recipients follow-up visits will occur at one month, 3 month, 6 months and 1 year post FMT.

Baseline stool samples will be collected from both the recipients and the UMMTP samples for baseline metagenomic sequencing. Recipient stool samples will be obtained weekly for the first month, then at 3 months, 6 months and 1 year. Microbiome analyses will also performed on recipient all stool samples post FMT to assess for successful engraftment of donor's microbiota onto the recipient's.

ELIGIBILITY:
Recipient Inclusion Criteria:

1. Age >18
2. One or more prior episode(s) of uncomplicated diverticulitis, as confirmed by imaging and clinical symptoms.
3. Eligible for surgical resection

Recipient Exclusion Criteria:

1. Subjects <18 years of age
2. Patients with active diverticulitis flare
3. Evidence of complicated diverticulitis (diverticulitis with abscess/phlegmon, bleeding, stricture, fistula or perforation) on imaging
4. Prior fecal transplant
5. Patients unable to provide informed consent
6. Pregnant and/or breastfeeding women
7. Prisoners
8. Students
9. Prior small or large bowel obstruction within the past year
10. Prior major gastrointestinal or intra-abdominal surgery
11. Any major illness or condition that may substantially increase risks to the recipient based on the investigator's judgment.
12. Sexually active women who adhere to natural family planning alone

Donor Inclusion Criteria:

1. Adult patients ≥18 years old
2. Colonoscopy screening as recommended by the American Cancer Society. However, it is to be noted that only recipients will undergo colonoscopy for receipt of FMT as part of the study, not donors. We will only ensure that the prospective donor follows the recommended guidelines for screening colonoscopy, which are to begin at the age of 45. If the donor does not meet such guidelines, s/he will not be allowed to proceed as a donor. If a donor is not yet eligible to undergo screening colonoscopy (i.e., younger than 45), this will not be required of him/her."
3. Able to provide informed consent

Donor Exclusion Criteria:

1. History of diverticulitis
2. Recent COVID-19 infection, confirmed or suspected exposure to COVD-19 within the past eight weeks. Such subjects will be excluded irrespective of negative COVID nasopharyngeal test.
3. Risk of infectious agent

   * Known exposure to HIV, syphilis, or viral hepatitis (within the previous 12 months)
   * High-risk sexual behaviors including sexual contact with anyone with HIV/AIDS or hepatitis, men who have sex with men, sex for drugs or money
   * Use of illicit intravenous (IV) drug use
   * Tattoo or body piercing within 6 months
   * Incarceration within previous 12 months
   * Known current communicable disease (e.g., COVID 19, Influenza, STDs, HIV/AIDS, Hepatitis B and C)
   * Risk factors for variant Creutzfeldt-Jacob disease to prevent potential transmission of abnormal/pathologic prions (cellular proteins), which are the basis of this disease.
   * Receipt of blood transfusion from country other than the United States of America (USA) and Canada in the previous 6 months
4. Individuals who are at a higher risk for colonization with multi-drug resistant organisms (MDRO):

   * Health care workers
   * Persons who have been hospitalized or discharged from long-term care facilities in the past 30 days
   * Persons who regularly attend outpatient medical or surgical clinics
   * Persons who have engaged in medical tourism in the past 30 days
5. Gastrointestinal comorbidities

   * History of inflammatory bowel disease
   * History of celiac disease
   * History of irritable bowel syndrome, idiopathic chronic constipation, or chronic diarrhea
   * History of gastrointestinal malignancy
6. Other

   * Antibiotic use within the preceding 90 days
   * Ingestion of a potential allergen (e.g., nuts) where recipient has a known allergy to this agent within the past 30 days
   * Systemic autoimmunity (e.g., multiple sclerosis, connective tissue disease)
   * Chronic pain syndromes (e.g., chronic fatigue syndrome, fibromyalgia)
   * Fever, defined as temperature of 100 F or 38.7C, on the day of stool donation. Potential donors will be allowed to re-screen within 1 week if febrile on the day of stool donation. .
   * Sexually active women who adhere to natural family planning alone as method of contraception
   * Prisoners
   * Students
   * Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Number of diverticular flares/attacks since FMT | 1 year
  After FMT, recipients/participants will be asked to report the number of diverticulitis episodes they have experienced since FMT
Number of emergency room visits and hospitalizations due to diverticulitis since FMT | 1 year
  After FMT, recipients/participants will be asked to report the number of times (if any) they presented to the emergency room or were hospitalized due to diverticulitis.
Number of courses of antibiotics required for the treatment of diverticulitis since FMT | 1 year
  After FMT, recipients/participants will be asked to report whether they required any antibiotics due to diverticulitis
Necessity for surgery | 1 year
  After FMT, recipients/participants will be asked to report whether they required surgery to treat diverticulitis

CONTACTS AND LOCATIONS:
Overall Officials: Justin A Maykel, MD, Principal Investigator — UMass Chan Medical School
Locations (1):
- UMASS Memorial Medical Center, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No